CLINICAL TRIAL: NCT03750305
Title: Evaluating the Effectiveness of Imagery Focussed Therapy in Patients Suffering From Bipolar Disorder: an Exploratory Trial
Brief Title: Evaluating the Effectiveness of Imagery Focussed Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University (Other)
Responsible Party: Principal Investigator, Karin van den Berg, Clinical Psychologist, PhD student Maastricht University, Maastricht University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMCT in BD
Record Dates: First submitted 2018-02-27; First posted 2018-11-23 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Intervention Model Description: Between groups, comparing Imagery-Focussed therapy with psychoeducation/TAU/within group, comparing baseline phase with treatment phase.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- psychoeducation/TAU (Active Comparator): TAU consists of psycho-education for a period of 12 weeks, consisting of 6 2-hour sessions. Psycho-education is offered in groups,
  Interventions: Other: TAU
- imCT intervention (Experimental): For a period of 12 weeks, 12 1-hour sessions of imagery-focused Cognitive Therapy delivered weekly by a trained therapists, divided in an in depth identification (4 sessions) of images followed by imagery interventions, (6 sessions) and a consolidation phase (2 sessions).
  Interventions: Other: imagery-focused Cognitive Therapy

INTERVENTIONS:
Other: imagery-focused Cognitive Therapy — In depth identification phase: Therapists and patient collaboratively map out difficulties and pinpoint a treatment focus.
  Imagery interventions: The imagery intervention consists of metacognitive imagery rescripting or promoting positive imagery or competing tasks (or a combination of these).
  Consolidation: Consist of fine tuning the strategies, relapse prevention using a video diary.
  Other Names: ImCT
  Arms: imCT intervention
Other: TAU — Psycho-education is offered in groups, using the format described by Honig (Postma, Honig, & van Gent, 2008).
  Other Names: Psychoeducation
  Arms: psychoeducation/TAU

SUMMARY:
This study explores the effectiveness of a brief Imagery-focussed Cognitive Therapy (imCT) compared to psychoeducation, regarded as treatment as usual for this patient population, in patients suffering from BD receiving mood stabilising medication. ImCT was successfully tested in a pilot study using a case series design. The investigators now elaborate on this study comparing effectiveness of the intervention to psychoeducation/TAU.

DETAILED DESCRIPTION:
Bipolar disorder (BD) is a severe mental health illness affecting 1.9% to 2.4% of the population and is associated with high inter episode distress, ongoing mood swings (mood variability), high suicide risks and high co-morbidity (especially anxiety). 50% of patients do not recover within one year, and only 25% of patients achieve full recovery of function, despite receiving the recommended lead intervention consisting of pharmacotherapy (mood stabilisers such as lithium). Added psychoeducation and cognitive behavioural interventions (CBT) have only modest effects. Overall there is consensus for the need to update CBT and increase its effectiveness, aimed at not only managing symptoms but also targeting perpetuating or precipitating factors influencing symptoms, especially mood variability.

Recent studies suggest that patients with BD experience more vivid, compelling and upsetting mental images compared to patients suffering from unipolar depression and healthy controls and that this may contribute to or even maintain their clinical difficulties. That is, imagery in experimental research has proven to have a stronger effect on mood changes than verbal cognitions. The amplified imagery vividness of patients suffering from BD might therefore precipitate or perpetuate their mood variability. In many other mental health problems imagery interventions as a stand-alone intervention, or added to regular CBT, are offered with the aim to decrease imagery vividness or modify/update appraisals of imagery. In BD patients such interventions, therefore, might also target important precipitating or perpetuating factors influencing their mood problems.

This study aims to assess the effectiveness of a brief Imagery-focussed Cognitive Therapy (imCT) compared to psychoeducation, regarded as treatment as usual for this patient population, in patients suffering from BD receiving mood stabilising medication. ImCT was successfully tested in a pilot study using a case series design. The investigators now elaborate on this study comparing effectiveness of the intervention to psychoeducation/TAU. The investigators hypothesise that (1a) mood variability (primary outcome variable) and (1b) symptoms of depression, mania and anxiety (secondary outcome variables) show stronger decreases in BD patients receiving imCT than in patients receiving psychoeducation/TAU. Moreover, (2) in the imCT group this effect is expected to be mediated by changes in imagery which is targeted during this intervention (target imagery). The investigators also hypothese that (3) imagery frequency and compellingness and vividness of imagery reduce more in the imCT group than in the group receiving psychoeducation/TAU. The primary outcome variable, mood variability, is calculated using daily mood measurements, during a 4-week baseline, during the invention and after the end of intervention until follow up at 16 weeks, in both imCT and psychoeducation/TAU. Most secondary outcome variables are assessed using weekly online questionnaires, pre-and post intervention and at 8 and 16 weeks follow-up, anxiety is calculated both weekly online and using daily measurements (see below).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-68
* Sufficient Dutch language ability to permit the assessment to be completed.
* Diagnosis of DB (I or II or NOS) according to DSM-5 (clinicians assessment).
* Willing to complete daily and weekly monitoring throughout the duration of the study.
* Successful completion of the daily monitoring in the 4 weeks active run-in phase.
* Willing to be randomised to either imCT or psychoeducation/TAU condition
* Can commit to attending 12 consecutive weekly sessions imCT or psychoeducation/TAU.

Exclusion Criteria:

* Learning difficulties, organic brain disease or severe neurological impairment.
* Current severe substance or alcohol misuse (clinicians assessment).
* Current manic episode as diagnosed by DSM-5
* Current active psychotic symptoms
* Presence of active suicidal risk as indicated by a score of 2 or more on item 12 (i.e. frequent thought and/or plans to end their life) of the QIDS (Rush et al., 2003) confirmed by convergent clinical opinion.
* Taking part in concurrent treatment studies investigating pharmacological or psychological treatment for BD.

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline Mood variability to follow up at 16 weeks after end of intervention | The ALS-18 is administered at T0, after 4 weeks baseline at T1, after the end of intervention (12 weeks in the ImCT condition, and 6 weeks in the psychoeducation condition) T2, 8 weeks after the end of intervention T3, and after 16 weeks follow up -T4.
  Mood variability is measured using the Affect Lability Score Short Version (ALS-18; Oliver & Simons, 2004). The ALS-18 is a self-report scale measuring lability in affect and consists of 18 items. Ratings are made on a 4-point scale with a maximum score of 72. Scores range from A= very characteristic of me (4 points), to D= very uncharacteristic of me (1 point).

SECONDARY OUTCOMES:
Change from baseline Level of depression to follow up at to follow up at 16 weeks | measured weekly throughout the duration of the study in both groups (32 weeks imCT and 26 weeks psychoeducation/TAU).
  - Level of depression, using the Quick Inventory of Depressive Symptoms (QIDS-SR) (Rush et al., 2003). The QIDS-SR is a 16-item self-report rating scale in which the nine DSM 5 symptoms of major depression are incorporated. Answers are rated on a four-point Likert scale (0-3).
Change from baseline level of mania to follow up at 16 weeks | measured weekly throughout the duration of the study in both groups ( 32 weeks imCT and 26 weekspsychoeducation/TAU).
  - Level of mania, using the Altman Self-Rating Mania Scale (ASRM-NL) (Altman, Hedekker, & Peterson, 1997). The ASRM-NL is a 5 item self-report instrument to measure severity of mania symptoms. Answers are rated on a 5-point Likert scale, where higher scores indicate higher levels of mania. Total score ranges from 0 to 20, with a cut off score of 5 or more indicating relapse into mania.
Change from baseline level of anxiety to follow up at 16 weeks | measured both daily and weekly throughout the duration of the study in both groups (32 weeks imCT and 26 weeks psychoeducation/TAU)
  - Level of anxiety, using the Beck Anxiety Inventory (BAI) (Osman, Barrios, Aukes, Osman, & Markway, 1993). The BAI is a 21-item self-report questionnaire used for measuring the severity of anxiety. Answers are rated on a 4-point Likert scale (0-3). Total scores range from o to 63, where scores of 22 or more indicate moderate anxiety, 36 or more concerning levels of anxiety.
Change from baseline level of hopelessness to follow up at 16 weeks follow up | measured at baseline (T0), after 4 weeks pre-intervention (T1), post-intervention after 6 weeks in the psychoeduc condition and 12 weeks in the ImCT condition (T2) and at follow up at 8 weeks (T3) and at 16 weeks (T4).
  participants rate their hopelessness using the Beck Hopelessness Scale (Beck, Brown, & Steer, 1997), The BHS is a 20 item self-report scale measuring three aspects of hopelessness: feelings about the future, motivation and expectations. The BHS demonstrates good internal consistency (alpha = .93) and has high reliability in psychiatric samples (Beck et al., 1997)
Change from baseline level of general functioning and coping to follow up at 16 weeks | Participants rate their level of functioning at baseline (T0), after 4 weeks pre-intervention (T1), post-intervention12 weeks in the ImCT condition and 6 weeks in the psychoeducation condition (T2) and at follow up at 8 weeks (T3) and at 16 weeks (T4).
  Participants rate their level of functioning using the Longitudinal Interval Follow up Evaluation - Range of Impaired Functioning Tool (Leon, et al., 1999). This is a brief scale for people suffering from affective disorders, measuring four different functional areas (employment, interpersonal relations, satisfaction and recreation) on a 5 point Likert scale (low rating imply higher functioning).
Change from baseline level of mood variability to follow up at 16 weeks | Daily measurements throughout the duration of the study, 32 weeks for the participants in the ImCT condition and 26 weeks for the participants in the psychoeducation condition
  Mood variability, using daily measurements of both mania and depression with the National Institute of Mental Health Life Chart Methodology (NIMH-LCM) Prospective Self-Rating (Denicoff et al., 2000; Leverich and Post, 1998). Participants rate their mood (both mania and depression) on a 11-point likert scale, ranging from -4 (severe depression, admission required due to severe dysfunction) to 0 (stable mood) to +4 (severe mania, admission required due to severe dysfunction).
Change from baseline level of anxiety to follow up at 16 weeks | Daily measurements throughout the duration of the study, 32 weeks for the participants in the ImCT condition and 26 weeks for the participants in the psychoeducation condition
  Anxiety is measured on a VAS scale indicating no anxiety (1) to severe anxiety (4).

OTHER OUTCOMES:
General Imagery (frequency of imagery, quality of imagery and appraisals of imagery): | administered at T0, after 4 weeks baseline at T1, after the end of intervention (12 weeks in the ImCT condition, and 6 weeks in the psychoeducation condition) T2, 8 weeks after the end of intervention T3, and after 16 weeks follow up -T4.
  This measured using a 42-item online Imagery Survey recently validated in a student sample, and presently used in an on-going current study comparing imagery aspects between patients suffering from BD, patients suffering from unipolar depression and imagery prone students without a present disorder. This is further assessed using the Mental Imagery and Coping with Bipolar Disorder Questionnaire (MICQ-BD) is a 14 item self-report instrument assessing patient's response to mental imagery on a five-point Likert scale, ranging from "not at all" to "a lot". In a pilot study Holmes (2016) calculated the internal conconsistency (alpha = .70) of this measure to be satisfactory (DiSimplicio et al., 2016).
Ratings of target imagery (moderator) | Measured weekly throughout the study for 32 weeks in the ImCT condition and 26 weeks in the psychoeducation condition
  Changes in target imagery are measured in order to test if reductions in moodvariablity compared to baseline (i.e. the primary objective) are mediated by reductions in levels of problematic imagery during treatment. The Visual Analogue Scales of Imagery Characteristics (VAS Imagery) have been tailored to BD population rating on a scale 0-9, for example such as: "How real / vivid / absorbing / preoccupying / compelling have your image(s) been over the past week'"; "To which extent could you understand the role that the image(s) play in your mood instability?"; "To which extent could you find positive / helpful way of using the image(s)?". Target imagery is measured weekly throughout the duration of the study in the imCT group.
General Imagery | administered at T0, after 4 weeks baseline at T1, after the end of intervention (12 weeks in the ImCT condition, and 6 weeks in the psychoeducation condition) T2, 8 weeks after the end of intervention T3, and after 16 weeks follow up -T4.
  Changes in general imagery are measured using the Mental Imagery and Coping with Bipolar Disorder Questionnaire (MICQ-BD) is a 14 item self-report instrument assessing patient's response to mental imagery on a five-point Likert scale, ranging from "not at all" to "a lot". In a pilot study Holmes (2016) calculated the internal conconsistency (alpha = .70) of this measure to be satisfactory (DiSimplicio et al., 2016).

CONTACTS AND LOCATIONS:
Overall Officials: karin van den Berg, Principal Investigator — Maastricht University
Locations (1):
- Centrum Bipolair, GGzE, Eindhoven, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van den Berg KC, Hendrickson AT, Hales SA, Voncken M, Keijsers GPJ. Comparing the effectiveness of imagery focussed cognitive therapy to group psychoeducation for patients with bipolar disorder: A randomised trial. J Affect Disord. 2023 Jan 1;320:691-700. doi: 10.1016/j.jad.2022.09.160. Epub 2022 Oct 5. PMID 36206888
- See also: Applications of time-series analysis to mood fluctuations in bipolar disorder to promote treatment innovation: a case series — https://www.ncbi.nlm.nih.gov/pubmed/26812041
- See also: An investigation of mental imagery in bipolar disorder: Exploring "the mind's eye". — https://www.ncbi.nlm.nih.gov/pubmed/27995690
- See also: Evidence-based guidelines for treating bipolar disorder Revised third edition recommendations from the British. — https://maastrichtuniversity.on.worldcat.org/oclc/6035584563
- See also: Mental imagery as an emotional amplifier: application to bipolar disorder — https://www.ncbi.nlm.nih.gov/pubmed/18990364

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-01): https://cdn.clinicaltrials.gov/large-docs/05/NCT03750305/Prot_SAP_000.pdf